CLINICAL TRIAL: NCT03097861
Title: A Randomized, Placebo-controlled, Double-blinded, Multicenter Study of the Bioequivalence of Sprinkle and Capsule Formulations of Lubiprostone, as Compared to Placebo, in Adult Subjects With Chronic Idiopathic Constipation
Brief Title: Evaluation of the Bioequivalence of Sprinkle and Capsule Formulations of Lubiprostone, as Compared to Placebo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sucampo Pharma Americas, LLC (Industry)
Collaborators: Sucampo AG (Industry); Sucampo Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCMP-0211-302
Record Dates: First submitted 2017-03-27; First posted 2017-03-31 (Actual); Results first posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Chronic Idiopathic Constipation
MeSH Terms: interventions — Lubiprostone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lubiprostone Capsule (Active Comparator): Lubiprostone 24 mcg capsule twice daily (BID) for 7 days.
  Interventions: Drug: Lubiprostone
- Lubiprostone Sprinkle (Experimental): Lubiprostone 24 mcg sprinkle BID for 7 days.
  Interventions: Drug: Lubiprostone
- Placebo (Placebo Comparator): Placebo matching to lubiprostone (sprinkle/capsule) BID for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lubiprostone — 24 mcg administered orally BID
  Other Names: Amitiza
  Arms: Lubiprostone Capsule; Lubiprostone Sprinkle
Drug: Placebo — 24 mcg administered orally BID
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the bioequivalence of sprinkle and capsule formulations of lubiprostone, as compared to placebo, when administered orally in participants with Chronic Idiopathic Constipation (CIC).

ELIGIBILITY:
Inclusion Criteria:

* Either has medically-confirmed diagnosis of chronic constipation (per Rome III), or meets the diagnosis as confirmed using the Rome III constipation module questionnaire during the Screening period.
* Is male or female, 18 or older years of age
* Should be on stable dose of fiber supplement or a concomitant medication for the indication of lowering blood pressure

Exclusion Criteria:

* Has any gastrointestinal (GI) condition, other than constipation, affecting GI motility or defecation
* Is unable to eat or drink, take oral medications, or to hold down oral medications due to vomiting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 552 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2017-08-17 (Actual); Study Completion 2017-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Mallinckrodt
Locations (63):
- United States (63):
  - Investigative Site, Birmingham, Alabama
  - Investigative Site, Foley, Alabama
  - Investigative Site, Little Rock, Arkansas
  - Investigative Site, Anaheim, California
  - Investigative Sitee, Chula Vista, California
  - Investigative Site, Garden Grove, California
  - Investigative Site, Long Beach, California
  - Investigative Site, Los Angeles, California
  - Investigative Site, Panorama City, California
  - Investigative Site, San Diego, California
  - Investigative Site, San Marcos, California
  - Investigative Site, Upland, California
  - Investigative Site, Colorado Springs, Colorado
  - Investigative Site, New London, Connecticut
  - Investigative Site, Clearwater, Florida
  - Investigative Site, Coral Springs, Florida
  - Investigative Site, DeLand, Florida
  - Investigative Site, Hialeah, Florida
  - Investigative Site, Jupiter, Florida
  - Investigative Site, Miami, Florida
  - Investigative Site 2, Miami, Florida
  - Investigative Site, Orlando, Florida
  - Investigative Site, Plantation, Florida
  - Investigative Sitee, Port Orange, Florida
  - Investigative Site, Port Saint Lucie, Florida
  - Investigative Site, Tampa, Florida
  - Investigative Site, West Palm Beach, Florida
  - Investigative Site, Athens, Georgia
  - Investigative Site, Snellville, Georgia
  - Investigative Site, Stockbridge, Georgia
  - Investigative Site, Blackfoot, Idaho
  - Investigative Site, Boise, Idaho
  - Investigative Site, Meridian, Idaho
  - Investigative Site, Lake Charles, Louisiana
  - Investigative Site, New Orleans, Louisiana
  - Investigative Site, Shreveport, Louisiana
  - Investigative Site, Chevy Chase, Maryland
  - Investigative Site, Hagerstown, Maryland
  - Investigative Site, New Bedford, Massachusetts
  - Investigative Site, Jackson, Missouri
  - Investigative Sitee, Bellevue, Nebraska
  - Investigative Site, Las Vegas, Nevada
  - Investigative Site, The Bronx, New York
  - Investigative Sitee, High Point, North Carolina
  - Investigative Site, Raleigh, North Carolina
  - Investigative Site, Cleveland, Ohio
  - Investigative Site, Mentor, Ohio
  - Investigative Site, Midwest City, Oklahoma
  - Investigative Site, Philadelphia, Pennsylvania
  - Investigative Site, Charleston, South Carolina
  - Investigative Site, Spartanburg, South Carolina
  - Investigative Site, Chattanooga, Tennessee
  - Investigative Site 2, Jackson, Tennessee
  - Investigative Site, Jackson, Tennessee
  - Investigative Site, Houston, Texas
  - Investigative Site, Longview, Texas
  - Investigative Site, McAllen, Texas
  - Investigative Site, Sugar Land, Texas
  - Investigative Site, Layton, Utah
  - Investigative Site, Taylorsville, Utah
  - Investigative Site, West Jordan, Utah
  - Investigative Site, Newport News, Virginia
  - Investigative Site, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adams A, Barish C, Chen A, Dennis P, Krause R, Lichtlen P, Losch-Beridon T, Mareya S, Schneider J. Capsule and Sprinkle Formulations of Lubiprostone Are Not Biologically Similar in Patients with Functional Constipation. Adv Ther. 2021 Jun;38(6):2936-2952. doi: 10.1007/s12325-021-01707-9. Epub 2021 Apr 8. PMID 33834354

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at 66 investigative sites in the United States.
Pre-assignment Details: Actual randomization ratio of sprinkle:placebo:capsule (2:1:1) was different than the planned randomization ratio (1:1:1)
Groups:
- Placebo: Placebo matching to lubiprostone (sprinkle/capsule) twice daily (BID) for 7 days.
- Lubiprostone Capsule: Lubiprostone 24 mcg capsule BID for 7 days.
Period: Overall Study
Arm/Group | Placebo | Lubiprostone Sprinkle | Lubiprostone Capsule
Started | 145 | 276 | 131
Safety Population (Randomized and took at least one dose of study drug, by treatment actually received) | 143 | 275 | 130
Modified Intent to Treat (As randomized, received at least one dose of study drug and had at least one diary entry) | 143 | 275 | 130
Completers (Completed the entire treatment period with a recorded primary endpoint) | 129 | 255 | 121
Per-protocol Population (PP) (Main population for efficacy analysis) | 126 | 234 | 113
Completed | 138 | 254 | 122
Not Completed | 7 | 22 | 9
Not completed — Adverse Event | 3 | 8 | 4
Not completed — Investigator Decision | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 7 | 1
Not completed — Withdrawal by Subject | 1 | 5 | 3
Not completed — Reason not provided | 3 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Per Protocol Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lubiprostone Sprinkle | Lubiprostone Capsule | Total
Number analyzed (Participants) | 126 | 234 | 113 | 473
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (13.32) | 47.4 (13.17) | 48.8 (13.38) | 47.6 (13.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 202 | 92 | 399
  Male | 21 | 32 | 21 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 64 | 33 | 128
  Not Hispanic or Latino | 95 | 170 | 80 | 345
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 2 | 3
  Asian | 3 | 12 | 3 | 18
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 1 | 4
  Black or African American | 50 | 99 | 48 | 197
  White | 71 | 120 | 59 | 250
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Observed Spontaneous Bowel Movement (SBM) Count Within 1 Week
Description: Observed SBM count was based on the observed data reported in the electronic daily diary for the actual number of SBMs during the 1-week treatment period.
Time Frame: during the 1-week treatment period
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: SBMs/week
Groups:
- Placebo: Matching placebo
- Lubiprostone Sprinkle: Lubiprostone 24 mcg sprinkle twice daily (BID) for 7 days.
Arm/Group | Placebo | Lubiprostone Sprinkle | Lubiprostone Capsule
Number analyzed (Participants) | 126 | 234 | 113
SBMs/week
  Baseline | 1.38 (0.692) | 1.37 (0.693) | 1.35 (0.720)
  Week 1 | 3.68 (2.164) | 4.82 (3.658) | 5.74 (3.786)
Statistical Analysis 1: Comparison: Placebo vs Lubiprostone Sprinkle; Test type: Other — Treatment p-value is from ANCOVA using SBM count as dependent variable, treatment as fixed effect and baseline count as random effect; p = 0.0020, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Lubiprostone Capsule; Treatment p-value is from ANCOVA using SBM count as dependent variable, treatment as fixed effect and baseline count as random effect; Test type: Other; p < 0.0001, ANCOVA

2. Secondary Outcome: Mean SBM Consistency Score Within 1 Week
Description: Stool consistency associated with SBMs was rated according to the 7-point Bristol Stool Form Scale (1-7) where 1 = Separate hard lumps, like nuts (hard to pass), 2 = Sausage-shaped but lumpy, 3 = Like a sausage but with cracks on the surface, 4 = Like a sausage or snake, smooth and soft, 5 = Soft blobs with clear-cut edges (passed easily), 6 = Fluffy pieces with ragged edges, a mushy stool, 7 = Watery, no solid pieces; entirely liquid. Scores in the mid-range of this scale indicate better stool consistency.
Time Frame: during the 1-week treatment period
Population: PP population. Number of participants analysed indicates participants who were evaluated for this outcome measure at each categorical time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Lubiprostone Sprinkle | Lubiprostone Capsule
Number analyzed (Participants) | 123 | 230 | 111
score on a scale
  Baseline: number analyzed (Participants) | 116 | 218 | 103
  Baseline | 2.47 (1.122) | 2.39 (1.211) | 2.28 (1.045)
  Week 1 | 3.43 (1.270) | 3.94 (1.516) | 4.22 (1.409)

3. Secondary Outcome: Mean SBM Straining Score Within 1 Week
Description: Bowel straining associated with SBMs was rated on a scale of 0-4 where 0 = Absent, 1 = Mild, 2 = Moderate, 3 = Severe, 4 = Very severe. Higher score indicates more straining, so a worse condition.
Time Frame: during the 1-week treatment period
Population: PP population. Number of participants analysed indicates participants who were evaluated for this outcome measure at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Lubiprostone Sprinkle | Lubiprostone Capsule
Number analyzed (Participants) | 126 | 234 | 113
score on a scale
  Baseline: number analyzed (Participants) | 116 | 218 | 111
  Baseline | 2.39 (0.739) | 2.31 (0.911) | 2.40 (0.892)
  Week 1: number analyzed (Participants) | 123 | 230 | 113
  Week 1 | 1.76 (0.871) | 1.45 (0.937) | 1.19 (0.917)

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence (including clinically significant changes in laboratory values or other clinical tests) experienced by a participant administered a pharmaceutical product regardless of causal relationship with the treatment. A TEAE is an episode which occur after the administration of the first dose of study medication and within 7 days after final dose.
Time Frame: From first dose of study medication to follow-up (up to 15 days)
Population: Safety population, defined as all randomized participants who took at least one dose of double-blinded study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lubiprostone Sprinkle | Lubiprostone Capsule
Number analyzed (Participants) | 143 | 275 | 130
Participants | 21 | 40 | 73

ADVERSE EVENTS:
Time Frame: from first dose of study medication through a 1-week follow-up (up to 15 days)
Description: Treatment-related Adverse Events (TRAEs) were any event with possible, probably, or definite relationship with the study medication, and with an onset date on or after the first dose of study medication and with an onset date no more than 7 days after the last dose of study medication. TRAEs were collected in the safety population, defined as all randomized participants who took at least one dose of double-blinded study medication.
Arm/Group | Placebo | Lubiprostone Sprinkle | Lubiprostone Capsule
All-Cause Mortality (participants affected / at risk) | 0/143 | 0/275 | 0/130
Serious Adverse Events (participants affected / at risk) | 0/143 | 0/275 | 0/130
Other Adverse Events (participants affected / at risk) | 15/143 | 50/275 | 29/130
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=143) | Lubiprostone Sprinkle (N=275) | Lubiprostone Capsule (N=130)
Diarrhea (Gastrointestinal disorders) | 4 | 22 | 13
Nausea (Gastrointestinal disorders) | 3 | 10 | 11
Abdominal pain (Gastrointestinal disorders) | 3 | 4 | 4
Vomiting (Gastrointestinal disorders) | 0 | 0 | 4
Headache (Nervous system disorders) | 5 | 17 | 4

LIMITATIONS AND CAVEATS:
Actual randomization ratio (2:1:1) was different than the planned ratio (1:1:1).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-06): https://cdn.clinicaltrials.gov/large-docs/61/NCT03097861/Prot_SAP_000.pdf